CLINICAL TRIAL: NCT00445198
Title: A Phase 1/2a Study Evaluating the Safety, Pharmacokinetics, and Efficacy of ABT-263 in Subjects With Small Cell Lung Cancer or Other Non-Hematological Malignancies
Brief Title: A Phase 1/2a Study of ABT-263 in Subjects With Small Cell Lung Cancer (SCLC) or Other Non-Hematological Malignancies
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: AbbVie (prior sponsor, Abbott) (Industry)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Organization: AbbVie (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: M06-822; 2006-003298-28 (EudraCT Number); NCT00929513 (obsolete NCT alias)
Record Dates: First submitted 2007-03-06; First posted 2007-03-08 (Estimated); Last update posted 2018-06-06 (Actual); Status verified 2013-01

CONDITIONS: Small Cell Lung Cancer; Small Cell Lung Carcinoma
Keywords: SCLC
MeSH Terms: conditions — Small Cell Lung Carcinoma | interventions — navitoclax

ARMS (1):
- Phase 1 and Phase 2a (Experimental)
  Interventions: Drug: ABT-263

INTERVENTIONS:
Drug: ABT-263 — Phase 1 dosing under two different schedules: 14 days on drug, 7 days off or continuous dosing.
  - 50 patients with SCLC and non-hematologic malignancies. Enrollment is closed in this arm of the study.
  Phase 2a dosing under two different schedules: 14 days on drug, 7 days off or continuous dosing.
  - 40 patients with SCLC

SUMMARY:
The Phase 1 portion of the study will evaluate the pharmacokinetic profile and safety of ABT-263 with the objective of defining the dose limiting toxicity and maximum tolerated dose. (This portion of the study is complete). The Phase 2a portion of the study will evaluate ABT-263 at the defined recommended Phase 2 dose to obtain additional safety information and a preliminary assessment of efficacy.

ELIGIBILITY:
Inclusion Criteria:

* The subject must be >=18 years of age.(Phase 1 & 2a)
* Histologically and/or cytologically documented diagnosis of small cell lung cancer (North America & UK) or other non-hematological malignancy (North America only).(Phase 1 only)
* Histologically and/or cytologically documented diagnosis of SCLC.(Phase 2a)
* At least one prior chemotherapy treatment regimen(s) and their disease is refractory or experienced progressive disease following the treatment.(Phase 1)
* Extensive-stage SCLC & is chemotherapy naïve(US only) has experienced progressive disease following at least one chemotherapy regimen or their disease is refractory.(Phase 2a)
* Brain metastases with clinically controlled neurologic symptoms, defined as surgical excision and/or radiation therapy followed by 21 days of stable neurologic function & no evidence of CNS disease progression as determined by CT or MRI within 21 days prior to the first dose of study drug.
* ECOG performance score <= 2(Ph 1) <=1(Phase 2a)
* Must be receiving a stable dose of Selective Serotonin Reuptake Inhibitor (SSRI) anti-depressants 21 days prior to 1st dose of study drug.
* Adequate bone marrow, renal & hepatic function per local lab reference range at Screening as follows:

  * Bone marrow: Absolute Neutrophil count (ANC)>=1000/µL
  * Platelets>= 100,000/mm3
  * Hemoglobin>=9.0g/dL
  * Renal function: Serum creatinine<= 2.0mg/dL or calculated creatinine clearance>=50mL/min
  * Hepatic function&enzymes: AST and ALT<=3.0 x the upper normal limit(ULN) of institution's normal range
  * Bilirubin<=1.5xULN. If Gilbert's Syndrome may have Bilirubin> 1.5 x ULN
  * Coagulation: aPTT and PT<=1.2 x the upper limit of normal
* Should have archived diagnostic tissue available for assessment of Bcl-2 family protein expression.(Phase 2a)
* All female subjects not surgically sterile or postmenopausal(for at least 1 year)and non-vasectomized male subject must practice at least one method of birth control.

Exclusion Criteria:

* Underlying or predisposing condition of bleeding or currently exhibits signs of bleeding.
* Recent history of non-chemotherapy induced thrombocytopenia associated bleeding within 1 year prior to first dose of study drug.
* Active peptic ulcer disease or other potentially hemorrhagic esophagitis/gastritis.
* The subject has active immune thrombocytopenic purpura (ITP),active autoimmune hemolytic anemia (AIHA), or a history of being refractory to platelet transfusions (within 1 year prior to the first dose of study drug).
* Currently receiving or requires anticoagulation therapy or any drug or herbal supplements that affect platelet function, with exception of low-dose anticoagulation medications that are used to maintain the patency of a central intravenous catheter.
* Received any anti-cancer therapy including chemotherapy, immunotherapy, radiotherapy, hormonal (with the exception of hormones for hypothyroidism or estrogen replacement therapy (ERT), anti estrogen analogs, agonists required to suppress serum testosterone levels), or any investigational therapy within 14 days prior to the first dose of study drug, or has not recovered to less than a grade 2 adverse effect(s) of the previous therapy.
* Received a biologic (G-CSF, GM-CSF or erythropoietin) within 28 days prior to the first dose of study drug.
* Steroid therapy for anti-neoplastic intent within seven days prior to the first dose of study drug.
* Has consumed grapefruit or grapefruit products within 3 days prior to the first dose of study drug.
* Significant history of cardiovascular disease, renal, neurologic, psychiatric, endocrinologic, metabolic, immunologic, or hepatic disease that in the opinion of the investigator would adversely affect his/her participating in this study.
* Positive for HIV
* A history of other active malignancies within the past 3 years prior to screening, with the exception of:

  * Adequately treated in situ carcinoma of the cervix uteri
  * Basal or squamous cell carcinoma of the skin
  * Previous malignancy confined and surgically resected with curative intent
* Evidence of other clinically significant uncontrolled condition(s) including, but not limited to:

  * Active systemic fungal infection
  * Diagnosis of fever and neutropenia within 1 week prior to study drug administration.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Actual)
Dates: Start 2007-04; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Safety assessment | Repeating sequence of 14 days on therapy and 7 days off or continuous dosing
Dose limiting toxicity determination | Repeating sequence of 14 days on therapy and 7 days off or continuous dosing
Maximum tolerated dose determination | Repeating sequence of 14 days on therapy and 7 days off or continuous dosing
Pharmacokinetic profile evaluation | Repeating sequence of 14 days on therapy and 7 days off or continuous dosing

SECONDARY OUTCOMES:
Extended safety assessment at the recommended Phase 2 dose | Repeating sequence of 14 days on therapy and 7 days off or continuous dosing
Preliminary efficacy assessment | Repeating sequence of 14 days on therapy and 7 days off or continuous dosing

CONTACTS AND LOCATIONS:
Locations (18):
- United States (14):
  - Site Reference ID/Investigator# 13605, Peoria, Arizona
  - Site Reference ID/Investigator# 5261, Phoenix, Arizona
  - Site Reference ID/Investigator# 11942, Los Angeles, California
  - Site Reference ID/Investigator# 4718, Sacramento, California
  - Site Reference ID/Investigator# 3755, Aurora, Colorado
  - Site Reference ID/Investigator# 8324, Atlanta, Georgia
  - Site Reference ID/Investigator# 2623, Chicago, Illinois
  - Site Reference ID/Investigator# 2625, Baltimore, Maryland
  - Site Reference ID/Investigator# 12343, Bethesda, Maryland
  - Site Reference ID/Investigator# 11941, Boston, Massachusetts
  - Site Reference ID/Investigator# 2626, Boston, Massachusetts
  - Site Reference ID/Investigator# 4934, Charlotte, North Carolina
  - Site Reference ID/Investigator# 2624, Nashville, Tennessee
  - Site Reference ID/Investigator# 6650, Tacoma, Washington
- Canada (2):
  - Site Reference ID/Investigator# 7493, Edmonton
  - Site Reference ID/Investigator# 7635, Ottawa
- United Kingdom (2):
  - Site Reference ID/Investigator# 18541, Leicester
  - Site Reference ID/Investigator# 2622, Manchester

REFERENCES:
- [Result] Gandhi L, Camidge DR, Ribeiro de Oliveira M, Bonomi P, Gandara D, Khaira D, Hann CL, McKeegan EM, Litvinovich E, Hemken PM, Dive C, Enschede SH, Nolan C, Chiu YL, Busman T, Xiong H, Krivoshik AP, Humerickhouse R, Shapiro GI, Rudin CM. Phase I study of Navitoclax (ABT-263), a novel Bcl-2 family inhibitor, in patients with small-cell lung cancer and other solid tumors. J Clin Oncol. 2011 Mar 1;29(7):909-16. doi: 10.1200/JCO.2010.31.6208. Epub 2011 Jan 31. PMID 21282543